CLINICAL TRIAL: NCT03196687
Title: Frequency of Asymptomatic Left Ventricular Diastolic Dysfunction in Diabetes Mellitus Type 2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mena samwel, Assiut University, Assiut University
Other Study IDs: assiut university9000
Record Dates: First submitted 2017-05-06; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-05

CONDITIONS: Diastolic Dysfunction
Keywords: diastolic dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with type 2 DM may develop a cardiomyopathy often called diabetic cardiomyopathy which is characterized by left ventricular diastolic dysfunction in early stages

Type 2 DM is associated with various types of subclinical target organ damage resulting in elevated risk of CVD events, moreover there is growing evidence that a prediabetic status, such as impaired fasting glucose is also related to subclinical target organ damage when compared to a group with normal glucose metabolism Diabetes mellitus is a well-studied major risk factor for coronary heart diseases, which is one of the leading causes of death worldwide. Another distinct entity of diabetes-related cardiac affection is the diabetic cardiomyopathy. This entity of cardic affection by diabetes still needs more and more attention, not only because it is common in diabetic patients, but also because of its easy detection by the simple, inexpensive and widely available diagnostic echocardiography.

DETAILED DESCRIPTION:
Patients with type 2 DM may develop a cardiomyopathy often called diabetic cardiomyopathy which is characterized by left ventricular diastolic dysfunction in early stages

Type 2 DM is associated with various types of subclinical target organ damage resulting in elevated risk of CVD events, moreover there is growing evidence that a prediabetic status, such as impaired fasting glucose is also related to subclinical target organ damage when compared to a group with normal glucose metabolism

Diabetes mellitus is a well-studied major risk factor for coronary heart diseases, which is one of the leading causes of death worldwide. Another distinct entity of diabetes-related cardiac affection is the diabetic cardiomyopathy. This entity of cardic affection by diabetes still needs more and more attention, not only because it is common in diabetic patients, but also because of its easy detection by the simple, inexpensive and widely available diagnostic echocardiography.

The proposed mechanisms that may be implicated in the pathogenesis of diabetic cardiomyopathy include autonomic dysfunction, microvascular disease, interstitial fibrosis and metabolic disorders. However, the actual causes and mechanisms remain unclear.

ELIGIBILITY:
Inclusion Criteria:

* DM type 2 who are asymptomatic of any cardiac symptom.

Exclusion Criteria:

* Patients of known hypertension with or without treatment.
* Cardiac arrhythmias.
* Cardiomyopathy.
* Valvular heart disease.
* Heart failure.
* Chronic pulmonary disease.
* Extreme age.
* Chronic renal failure.
* Subjects with poor transthoracic echo window.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Will assess the prevelance and frequency of diastolic dysfunction of the left ventricle in patients with asymptomatic type 2 DM and to explore its relation to other parameters, including patients' age, sex, the duration of diabetes and glycemic control.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
percentage of Frequency of asymptomatic left ventricular diastolic dysfunction in diabetes mellitus type 2 | 1 year

IPD SHARING:
Plan to Share IPD: Undecided
This study will assess the prevelancea and frequency of diastolic dysfunction of the left ventricle in patients with asymptomatic type 2 DM and to explore its relation to other parameters, including patients' age, sex, the duration of diabetes and glycemic control.